CLINICAL TRIAL: NCT06741202
Title: Recovery-oriented Group Therapy for Veteran Men With Military Sexual Trauma (CDA 23-054)
Brief Title: Recovery-oriented Group Therapy for Veteran Men With Military Sexual Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDX 24-005; IK2HX003783-01A2 (NIH)
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sexual Trauma
Keywords: military sexual trauma; veteran men; group therapy
MeSH Terms: conditions — Sexual Trauma; Military Sexual Trauma

STUDY DESIGN:
Intervention Model Description: Conduct a pilot randomized controlled trial with men MST survivors (n=32), randomized to the MMG or Present-Centered Group Therapy (PCGT; control condition) (four cohorts: 2 experimental, 2 control). Investigate engagement (session attendance) as well as recovery-oriented outcomes (agency, hope, belongingness, shame-reduction) and psychological symptoms (PTSD, MDD, suicidality) assessed at pre-, immediate post-, and 6-month post-intervention.
Who Masked: Participant
Masking Description: Participants will be allocated to either MMG or PCGT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Men's MST Group (MMG) (Experimental): This is a 12-week long group that meets for 90 minutes weekly. This group will draw on interventions, developed in our pilot study, and also based on the PI's previous clinical experience designing and delivering a men's MST Group oriented to reduce psychiatric distress including identity-based shame by promoting group discussion among Veteran men about masculinity, sexuality, belongingness, and emotion regulation. The group is oriented around building core drivers of recovery: 1) agency through exposure- and mindfulness-based interventions to improve distress management; 2) social belongingness through group discussions on gender-specific themes; and 3) hope through coping skill training and treatment experienced as relevant. The protocol will be further revised based on research activity during Aims 1 and 2.
  Interventions: Behavioral: Men's MST Group
- Present-Centered Group Therapy (PCGT) (Active Comparator): PCGT is a time-limited treatment for PTSD that focuses on increasing adaptive responses to current life stressors and difficulties that are directly or indirectly related to trauma or PTSD symptoms. PCGT was initially developed as a nonspecific comparison condition to test the effectiveness of trauma-focused cognitive behavioral therapy. The number of PCGT sessions has ranged from 12 to 32 for the group format, and is thus appropriate to utilize for the nature of this study. To minimize possible confounds, PCGT will be delivered for a 12-week period. The basis of PCGT is to provide "common factors" of psychotherapy, demonstrating the effects of what is unique in therapies. In this instance, PCGT may help articulate whether the effect of MMG is due to being gender-specific (bringing men together in the same group therapy setting) or being gender-tailored (delivering treatment that is specifically oriented to men, such as MMG group discussions).
  Interventions: Behavioral: Present-Centered Group Therapy

INTERVENTIONS:
Behavioral: Men's MST Group — see above
  Arms: Men's MST Group (MMG)
Behavioral: Present-Centered Group Therapy — see above
  Arms: Present-Centered Group Therapy (PCGT)

SUMMARY:
VA has identified military sexual trauma (MST) as one of its highest priorities. MST is associated with increased prevalence of PTSD and depression, substance use disorders, suicide, difficulties maintaining relationships and employment, and homelessness. Yet important gender differences have been identified among MST survivors and many man may experience stigma and shame related to masculinity and sexuality. While gender-based shame appears central to MST-related distress and treatment underutilization, gender has often been overlooked in establishing evidence-based approaches, and no VA MST-related treatment has been developed specifically for men. To address this critical service gap, this study will collect data on improving treatment strategies and patient engagement for men with histories of MST. It will seek to develop strategies for enhancing a 12-session, gender-tailored group therapy for men MST survivors previously developed and implemented by the principal investigator. It will interview Veteran participants and mental health clinicians, conduct a pilot randomized trial, and evaluate feasibility within the VA, with the long-term goal of national implementation

DETAILED DESCRIPTION:
Approximately 3.5% of Veteran men and 44% of Veteran women report a history of military sexual trauma (MST).Although women disproportionately experience MST, the absolute number of men who report MST (55,500 from 2004-2013) is relatively similar due to the larger proportion of men in the military. Further, MST likely remains vastly underreported among men, who experience multiple barriers to disclosure. Men survivors often wait decades to seek care for MST-related distress, contributing to pervasive life impairment.

MST is associated with transdiagnostic complexity and is associated with increased prevalence of PTSD and depression, substance use disorders, suicide, difficulties maintaining relationships and employment, and homelessness. Important gender differences have been identified among MST survivors: men may experience stigma and shame related to masculinity and sexuality; the probability of opioid use disorder among men with a history of MST is nearly double that of women; and men with histories of MST also experience more severe PTSD symptoms, chronic mental health symptoms, sexual dysfunction and distress, and greater risk for homelessness. While gender-based shame appears central to MST-related distress and treatment underutilization, gender has often been overlooked in establishing evidence-based approaches, and no VA MST-related treatment has been developed specifically for men.

To address this critical service gap, I designed a 12-session, gender-tailored, multi-modal, recovery-oriented group therapy for men MST survivors as part of my clinical responsibilities as a VA staff psychologist. My intervention (the Men's MST Group, or MMG), which I have been delivering continuously for 5 years, is based on the Integrated Recovery-oriented Model (IRM) for mental health services, and promotes agency through delivery of dynamic, exposure- and mindfulness-based techniques intended to improve distress management, social belongingness, and hope. This transdiagnostic intervention also seeks to reduce shame. Exploratory evaluation signaled strong retention, as well as recovery and attitudinal shifts, including reductions in shame and PTSD symptoms. As one participant noted after completing the MMG, "I can say the word 'rape' without shame." Given these initial findings, rigorous research is warranted to refine, test, and prepare for implementation of the intervention. Moreover, given the fact that most participants wait decades to seek treatment, more research is needed to facilitate men's utilization of MST-related services. In this proposed CDA, guided by Intervention Mapping and the Access Re-conceptualization Model, I plan to iteratively refine the MMG by interviewing Veteran participants and mental health clinicians, conducting a pilot randomized trial, and evaluating feasibility within the VA, with the long-term goal of national implementation.

This mentored CDA will fill gaps in my training - particularly in gender-tailored intervention development, intersectionality, clinical trials and health services research, and mixed methods - to support my independence as a VA clinician scientist focused on enhancing mental health services for vulnerable Veteran populations. The Specific Aims are to:

Aim 1. Revise the MMG treatment protocol, with attention to factors that will support men's access to, and engagement and retention in, mental health interventions. 1a) Conduct semi-structured qualitative interviews (n=24) with VA mental health clinicians, Vet Center clinicians, MST coordinators, and MST experts. Findings will inform protocol revisions. 1b) Review the revised protocol by conducting two focus groups with the two recent MMG cohorts (n=8). 1c) Convene an Expert Panel with selected Aim 1a participants and VA Operations Partners to finalize the protocol.

Aim 2. Using the revised protocol, conduct a pilot randomized controlled trial (RCT) with men MST survivors (n=32), randomized to the MMG or Present-Centered Group Therapy (PCGT; control condition) (four cohorts: 2 experimental, 2 control). Investigate engagement (session attendance) as well as recovery-oriented outcomes (agency, hope, belongingness, shame-reduction) and psychological symptoms (PTSD, MDD, suicidality) assessed at pre-, immediate post-, and 6-month post-intervention.

Aim 3. Assess pilot RCT findings and plan for multisite trial (Year 5 Merit). 3a) Conduct post-intervention semi-structured interviews with RCT participants and interventionists to understand treatment engagement factors as well as perceptions of accessibility, feasibility, acceptability, appropriateness, and effectiveness. 3b) Reconvene the Aim 1c Expert Panel to discuss RCT results and potential facilitators, barriers, and strategies for implementation of the MMG in usual VA mental health care. 3c) In collaboration with operations partners, enhance the protocol and design the intervention package with system-level considerations in preparation for a multisite trial.

VA has identified MST as one of its highest priorities. Given the prevalence of MST among men and the deleterious, often protracted MST-related symptomatology, it is critical to develop tailored services for this population. This application responds to VA HSR&D's research priorities of suicide prevention, mental health, and health equity, and ORD's priorities of increasing the real-world impact of VA research and actively promoting equity.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include any individual who identifies as a Veteran cisgender man with a history of MST, English-speaking, 18 years of age or older, and enrolled in the VAGLA. Participants must:

  * comprehend and sign the informed consent form
  * report a history of MST
  * agree to complete research instruments
* Because we are looking for a range of impact among men MST survivors, participants will not be excluded based on psychiatric diagnosis

Exclusion Criteria:

* Per chart review conducted by the PI prior to screening and patient contact, Veterans will be excluded if they demonstrate:

  * severe suicidal or homicidal ideation, defined using the Columbia Suicide Severity Rating Scale (C-SSRS) and behavioral flags per chart review
  * severe and uncontrolled substance abuse (identified through current treatment of a substance use disorder in chart)
  * illness that inhibits engagement in study procedures (e.g., inability to attend in-person visits)
  * inability to self-consent to participate
  * completion of CPT, PE, or the MMG 5 or fewer years ago
  * concurrent enrollment in a trauma-focused intervention
* Through chart review, Veterans who dropped out of these treatments after 3 sessions will still be eligible as this is considered "early dropout."
* If immediate clinical attention is warranted, Veterans will receive immediate care via procedures outlined in the human subjects protection plan

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — this is a study on men's MST
Enrollment: 32 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The Recovery Assessment Scale | up to 9 months
  The Recovery Assessment Scale (RAS) is a 41-question forced choice 5-level Likert rating scale, designed to assess recovery, with emphasis on agency, hope, and belongingness, and shame-reduction-key constructs postulated to impact and be expressive of psychological distress and intra- and inter-personal avoidance.The RAS is the most widely used instrument to measure recovery and has good internal consistency, test-retest reliability, and interrater reliability. The scale ranges with a minimum score of 24 and a maximum score of 120; higher values signifying higher recovery.
External and Internal Shame Scale | up to 9 months
  External and Internal Shame Scale (EISS) assesses global shame experience, with attention to its external and internal dimensions, relevant to men's MST. The scale consists of eight items, and measures four central shame domains: inferiority/inadequacy, sense of exclusion, uselessness/emptiness and criticism/judgment. This scale is found to have internal consistency and concurrent validity. The scale ranges with a minimum score of 0 and a maximum score of 32; higher values signifying higher levels of shame.
General Belongingness Scale | up to 9 months
  General Belongingness Scale (GBS), a 12-item measure rated on a 7-point Likert scale, assesses a general sense of belonging, another indication of interpersonal distress pertaining to MST. This scale is a reliable and valid brief measure of general belongingness, and shows good cross-cultural validity. The scale ranges with a minimum score of 0 and a maximum score of 72; higher values signifying higher levels of belongingness.

SECONDARY OUTCOMES:
Post-Traumatic Checklist for The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) | up to 9 months
  The PCL-5 is a 20-item non-MST specific self-report measure that assesses the DSM-5 symptoms of PTSD, a common indicator of MST-related distress. Each symptom is rated on a 5-point Likert scale assessing distress of each symptom. The PCL-5 has high reliability and validity, and provides a total and cluster symptom severity score corresponding with DSM-5 diagnostic criteria. The scale ranges with a minimum score of 0 and a maximum score of 80; higher values signifying higher levels of post-traumatic stress.
Patient Health Questionnaire-9 | up to 9 months
  Patient Health Questionnaire-9 (PHQ-9) is a widely used brief, 9-item instrument for screening, diagnosing, monitoring, and measuring the severity of depression over the course of two weeks. The PHQ-9 is a reliable and valid measure of depression severity that assess DSM criteria of depression, including suicidality. PHQ-9 has high cross-cultural validity and is often used in health care research. The scale ranges with a minimum score of 0 and a maximum score of 27; higher values signifying higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Yahalom, PhD MA, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No